CLINICAL TRIAL: NCT07066514
Title: Effectiveness of Exercises Supervised Via an Artificial Intelligence-Supported Mobile Application in Patients With Knee Osteoarthritis
Brief Title: Effectiveness of AI-Supervised Mobile Exercise Application in Patients With Knee Osteoarthritis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Selim Mahmut GÜNAY, Asst Prof, Mustafa Kemal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025-2/19
Record Dates: First submitted 2025-07-04; First posted 2025-07-15 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI-Based Mobile Home Exercise Group (Experimental)
  Interventions: Behavioral: AI-Supervised Mobile Exercise Program
- Standard Home Exercise Group (Experimental)
  Interventions: Behavioral: Booklet-Guided Home Exercise Program

INTERVENTIONS:
Behavioral: AI-Supervised Mobile Exercise Program — This intervention involves the use of an artificial intelligence (AI)-supported mobile application that delivers a personalized exercise program to patients with knee osteoarthritis. The app supervises exercise execution in real time using the device's camera and AI algorithms to track movements, count repetitions, and assess form accuracy. The program includes stretching, strengthening, and range of motion exercises performed 3-4 times per week for 4 weeks. The app provides instructional videos, personalized feedback, reminders, and records user performance. No video or personal images are stored; only anonymized motion data are collected and securely stored.
  Arms: AI-Based Mobile Home Exercise Group
Behavioral: Booklet-Guided Home Exercise Program — This intervention provides patients with a standardized home exercise program in printed booklet format. The program includes the same evidence-based stretching, strengthening, and range of motion exercises used in the mobile application group, performed 3-4 times per week for 4 weeks. Participants receive one-time in-person instruction on proper form but no ongoing supervision or feedback during the program. Adherence and technique are self-monitored.
  Arms: Standard Home Exercise Group

SUMMARY:
This study aims to evaluate the effectiveness of an artificial intelligence (AI)-supported mobile application that supervises home-based exercise programs in patients with knee osteoarthritis. A total of 80 participants aged 40 to 80 will be randomly assigned to one of two groups: a mobile application exercise group or a home exercise booklet group. Both groups will receive the same standardized stretching, strengthening, and range of motion exercises designed for knee osteoarthritis. The mobile app provides real-time feedback and supervision using the device's camera and artificial intelligence algorithms to track and guide exercise performance.

Participants in the app group will perform exercises with supervision via the app interface, while the control group will follow the same exercises using printed instructions. Both groups will exercise 3 to 4 times per week for 4 weeks. The study will compare pain levels, physical function, and balance before and after the intervention using validated outcome measures such as the WOMAC Index and the Visual Analog Scale.

This study may help determine whether AI-supported digital tools can improve exercise adherence and outcomes in patients with knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 40 and 80 years
* Diagnosed with knee osteoarthritis according to ACR criteria
* Referred to physical therapy by a physician for knee osteoarthritis
* Able to use a smartphone or tablet
* Having regular access to the internet
* Voluntarily agrees to participate in the study

Exclusion Criteria:

* History of knee surgery or currently undergoing surgical treatment
* Received physical therapy or rehabilitation for knee OA within the past 6 months
* Lack of access to a mobile device or internet
* Any neurological, cardiovascular, or musculoskeletal condition that prevents safe participation in exercise
* Cognitive impairment or psychiatric disorder interfering with exercise adherence
* Inability to follow instructions or use the mobile app interface
* Any condition that would contraindicate participation in a home-based exercise program

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Baseline and Week 4
  The WOMAC is a validated questionnaire used to assess pain, stiffness, and physical function in patients with knee osteoarthritis. It consists of 24 items: 5 for pain, 2 for stiffness, and 17 for physical function. Each item is scored on a 5-point Likert scale (0 = none to 4 = extreme), with a total score range of 0 to 96. Higher scores indicate worse symptoms.
Visual Analog Scale (VAS) | Baseline and Week 4
  Change in pain severity measured by the Visual Analog Scale (VAS; range: 0-10; higher scores indicate worse pain) at baseline and at 6 weeks.
Timed Up and Go (TUG) Test | Baseline and Week 4
Functional Reach Test (FRT) | Baseline and Week 4
Single-Leg Stance Test | Baseline and Week 4
Exercise Execution Accuracy Assessed by Mobile Application | Before and during the 4-week intervention
  Accuracy of exercise adherence detection by the AI algorithm compared to physiotherapist assessment (% agreement)

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa Uludag University, Bursa, Nilüfer, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nelligan RK, Hinman RS, Kasza J, Crofts SJC, Bennell KL. Effects of a Self-directed Web-Based Strengthening Exercise and Physical Activity Program Supported by Automated Text Messages for People With Knee Osteoarthritis: A Randomized Clinical Trial. JAMA Intern Med. 2021 Jun 1;181(6):776-785. doi: 10.1001/jamainternmed.2021.0991. PMID 33843948
- [Background] Xiang XN, Wang ZZ, Hu J, Zhang JY, Li K, Chen QX, Xu FS, Zhang YW, He HC, He CQ, Zhu SY. Telehealth-Supported Exercise or Physical Activity Programs for Knee Osteoarthritis: Systematic Review and Meta-Analysis. J Med Internet Res. 2024 Aug 2;26:e54876. doi: 10.2196/54876. PMID 39094114